CLINICAL TRIAL: NCT03467724
Title: Clinical Evaluation of the Safety and Performance of Fractional RF for the Treatment of Surgical Scars Following Breast Augmentation, Abdominoplasty or Face Lift
Brief Title: Treatment of Surgical Scars Following Breast Augmentation, Abdominoplasty or Face Lift
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Venus Concept (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CS0717
Record Dates: First submitted 2018-02-14; First posted 2018-03-16 (Actual); Results first posted 2024-07-29 (Actual); Last update posted 2024-07-29 (Actual); Status verified 2024-02

CONDITIONS: Surgical Scar; Breast Augmentation; Abdominoplasty; Face Lift
Keywords: Fractional Radiofrequency

STUDY DESIGN:
Intervention Model Description: The subject will act as their own control. Each surgical scar will be compared at the 12-month follow-up to the pre-treatment baseline.
Masking Description: The blinded reviewer will review the baseline photographs of the surgical scar(s) and compare them to the photographs taken at follow-up Month 12.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Fractional radiofrequency (FRF) (Experimental): Subjects received 3 FRF treatments (monthly) over their scar following breast augmentation, abdominoplasty or face lift surgery.
  Interventions: Device: Fractional Radiofrequency (FRF)

INTERVENTIONS:
Device: Fractional Radiofrequency (FRF) — Fractional radiofrequency will be delivered to the area of the surgical scar.

SUMMARY:
Evaluator-blinded study of the safety and performance of fractional radiofrequency (FRF) for the treatment of surgical scars following breast augmentation, abdominoplasty or facelift. The study will enroll up to 50 female subjects requesting treatment of surgical scars following breast augmentation or abdominoplasty and up to 25 male and female subjects requesting treatment of surgical scars following facelift surgery. Subjects will receive a total of 3 treatments of their surgical scars at 1-month intervals. Subjects will be followed up at 10 months after their last treatment (12 months after the first treatment).

ELIGIBILITY:
Inclusion Criteria:

1. Healthy, female, subjects 20-60 years of age who are seeking treatment for their breast augmentation or abdominoplasty surgical scars or male and female patients 40-75 years of age who are seeking treatment for their face lift surgical scars.
2. A minimum of four weeks since surgery.
3. Able to read, understand and voluntarily provide written Informed Consent.
4. Able and willing to comply with the treatment/follow-up schedule and requirements.
5. Willing to avoid direct sunlight for the duration of the study.
6. Women of child-bearing age are required to be using a reliable method of birth control at least 3 months prior to study enrollment and for the duration of the study, and have a negative Urine Pregnancy test at baseline.

Exclusion Criteria:

* 1. Fitzpatrick skin types 5-6. 2. Implantable defibrillators, cardiac pacemakers, and other metal implants 3. Subjects with any implantable metal device in the treatment area 4. Pacemaker or internal defibrillator, or any other active electrical implant anywhere in the body (e.g. cochlear implant).

  5. Permanent implant in the treated area, such as metal plates and screws, or an injected chemical substance.

  6. Current or history of any kind of cancer, or pre-malignant moles. 7. Severe concurrent conditions, such as cardiac disorders. 8. Pregnancy or intending to become pregnant during the study and nursing. 9. Impaired immune system due to immunosuppressive diseases, such as AIDS and HIV, or use of immunosuppressive medications.

  10. History of diseases stimulated by heat, such as recurrent herpes simplex in the treatment area; may be enrolled only following a prophylactic regime.

  11. Poorly controlled endocrine disorders, such as diabetes. 12. Any active condition in the treatment area, such as sores, psoriasis, eczema, and rash.

  13. History of skin disorders, such as keloids, abnormal wound healing, as well as very dry and fragile skin.

  14. History of bleeding coagulopathies, or use of anticoagulants. 15. Use of isotretinoin (Accutane®) within six months prior to treatment. 16. Treating over tattoo or permanent makeup. 17. Excessively tanned skin from sun, tanning beds or tanning creams within the last two weeks.

  18. As per the practitioner's discretion, refrain from treating any condition which might make it unsafe for the patient.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female subjects are eligible for surgical scar treatment following breast augmentation and abdominoplasty. Both men and women are eligible for facelift scar treatments.
Enrollment: 54 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2020-04-13 (Actual); Study Completion 2020-04-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kai O. Kaye, Principal Investigator — Ocean Clinic
Locations (1):
- Ocean Clinic, Marbella, Spain

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 3 subjects failed screening and were not treated in the study.
Groups:
- FRF Treatment: Each subject received 3 VivaMD treatments (monthly).
Period: Overall Study
Arm/Group | FRF Treatment
Started | 51
Completed | 43
Not Completed | 8
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 1
Not completed — Protocol Violation | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Arm/Group | FRF Treatment
Number analyzed (Participants) | 51
Age, Continuous [Mean (Standard Deviation); unit: years] | 47.5 (0.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Mediterranean | 19
  Eastern European | 5
  Western European | 22
  Brazilian (White&Black) | 1
  Black | 1
  Central & South American | 2
  Iranian | 1

OUTCOME MEASURES:

1. Primary Outcome: Improvement of Surgical Scars at 12 Months Compared to Baseline (Pre-treatment) as Evaluated by 3 Independent Blinded Reviewers Using the General Aesthetic Improvement Scale (GAIS). The GAIS Ranges From 3 (Very Much Improved) to -3 (Very Much Worse).
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FRF Treatment
Number analyzed (Participants) | 43
units on a scale | 1.66 (0.71)

2. Secondary Outcome: Assessment of Surgical Scars at 12 Months as Evaluated by the Patients.
Description: Patient and Observer Scar Assessment Scale (POSAS) was used to evaluate the scar for pain, itching, color, stiffness, thickness, and appearance compared to their normal skin using a numbered scale. The scale ranges from 7 (no scar) to 70 with higher scores being worse and suggesting a worse scar.
Time Frame: 12 months
Measure: Mean (Standard Error); unit: units on a scale
Groups:
- 10 Months After FRF Treatment: Each subject received 3 VivaMD treatments (monthly).
- Baseline: Before treatment
Arm/Group | 10 Months After FRF Treatment | Baseline
Number analyzed (Participants) | 43 | 43
units on a scale | 13.4 (1.2) | 28.3 (1.4)

3. Secondary Outcome: Subject Satisfaction With Treatment
Description: Subjects will use the 5-point Likert Satisfaction scale where 4 is very satisfied, 3 is satisfied, 2 is having no opinion, 1 is unsatisfied and 0 is very unsatisfied to evaluate their satisfaction with the treatment.
Time Frame: 12 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | FRF Treatment
Number analyzed (Participants) | 43
units on a scale | 3.4 (1.0)

ADVERSE EVENTS:
Time Frame: 10 months
Arm/Group | FRF Treatment
All-Cause Mortality (participants affected / at risk) | 0/51
Serious Adverse Events (participants affected / at risk) | 0/51
Other Adverse Events (participants affected / at risk) | 3/51
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | FRF Treatment (N=51)
Wound Healing Disorder (post-op) (Skin and subcutaneous tissue disorders) | 2 (2)
Enlargement of Scar (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-02-07): https://cdn.clinicaltrials.gov/large-docs/24/NCT03467724/Prot_SAP_003.pdf